CLINICAL TRIAL: NCT05676268
Title: Clinical and Radiographic Outcomes of Implant-supported Full-ceramic Partial Fixed Dental Prostheses With Cantilever Extension: A Proof of Principle Study With a Follow-up of at Least 1 Year
Brief Title: Implant-supported Fixed Dental Prostheses (FDPs) With Cantilever Extension
Status: Completed | Type: Observational
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Other Study IDs: FDPs with cantilever
Record Dates: First submitted 2022-12-22; First posted 2023-01-09 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Dental Implant Failed; Prosthesis Failure; Peri-Implantitis
MeSH Terms: conditions — Prosthesis Failure; Peri-Implantitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with oral implants supporting full ceramic fixed dental prostheses
  Interventions: Procedure: Implant-supported fixed dental prostheses with cantilever extension

INTERVENTIONS:
Procedure: Implant-supported fixed dental prostheses with cantilever extension — Healthy patients in need of replacement of missing teeth with dental implants supporting partial fixed dental prostheses with cantilever extensions

SUMMARY:
To report the clinical and radiographic outcomes of implant-supported fixed dental prostheses with full-ceramic cantilever extensions (FDPCs) after a function time ≥ 12 months.

DETAILED DESCRIPTION:
Patients with full ceramic FDPCs in anterior and posterior areas will be clinically and radiographically re-evaluated. Mesial and distal radiographic marginal bone levels (mBLs) from baseline (i.e. delivery of FDPC) to the follow-up examination were calculated and compared between implant surfaces adjacent to and distant from the cantilever extension. Implant survival rate (%), pocket probing depth (PPD), presence/ absence of bleeding on probing (BoP) and presence/absence of mechanical/technical and biological complications were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years
* Written informed consent
* Patients with systemic health or controlled medical conditions
* Patients with healthy or treated periodontal conditions
* Patients enrolled in regular supportive periodontal therapy (SPT)
* Patients without clinical signs of bruxism and/or oral parafunctions
* 2 osseointegrated dental implants in the canine or posterior areas of maxilla and mandible following transmucosal placement and healing of 3-6 months
* Tissue level solid-screw implants with a sand-blasted and acid- etched (SLA) surface with an endosseous diameter of 3.3, 4.1 or 4.8 mm, a length of 8, 10 or 12 mm, a shoulder diameter of 4.8 mm and a supracrestal machined neck with a height of 1.8 or 2.8 mm (Straumann® Dental Implant System, Institut Straumann AG, Basel, Switzerland)
* Full-ceramic
* Utilization of prefabricated titanium abutments
* Cemented (3M™ ESPE Ketac™ Cem, Seefeld, Germany) or screw-retained fixed dental prostheses with a mesial or distal cantilever extension (FDPCs)
* Cantilever extension corresponding to 1 premolar unit (i.e., 6-7 mm)
* Absence of occlusal contacts or guidance on the cantilever extension at baseline
* Opposing dentition consisting of natural teeth or fixed or removable prosthetic restorations
* Availability of a periapical radiograph at baseline (i.e. FDPC delivery)
* Availability of PPD measurements (mm) taken at baseline at 4 sites/implant with a graduated Michigan periodontal probe (Deppeler SA, Rolle, Switzerland)
* Availability of BoP measurements (%) (Lang et al., 1986) taken at baseline at 4 sites/implant with a graduated Michigan periodontal probe (Deppeler SA, Rolle, Switzerland).

Exclusion Criteria:

* Untreated or active periodontal diseases
* Immediate implant placement (i.e., Type I implant placement according to Hämmerle et al., 2004)
* FDPCs in the aesthetic zone (i.e., replacement of maxillary or mandibular incisors)
* FDPCs supported by hollow-screw and hollow-cylinder implants

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with missing teeth rehabilitated with dental implants supporting partial fixed dental prostheses with cantilever extensions
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Implant survival rate | 12 months
  Percentage of dental implants present at follow-up visit

SECONDARY OUTCOMES:
Peri-implant marginal bone level changes | 12 months
Number of technical complications | 12 months
Number of mechanical complications | 12 months
Number of Biological complications | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Roccuzzo, Principal Investigator — University of Bern
Locations (1):
- Department of Periodontology, University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No